CLINICAL TRIAL: NCT01785355
Title: Periodontal Disease, Inflammation, Nutritional Status And Anaemia Response To Erythropoietin In Chronic Haemodialyzed Patients - The Impact Of Treatment For Periodontal Disease
Brief Title: The Impact Of Periodontal Disease Treatment On The General Health Status In Chronic Haemodialyzed Patients
Acronym: PAROHEM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Anemia Working Group Romania (Other)
Responsible Party: Principal Investigator, Oana Slusanschi, DMD, Anemia Working Group Romania
Other Study IDs: 005; 00022 (Registry Identifier: Romanian Renal Registry)
Record Dates: First submitted 2013-01-29; First posted 2013-02-07 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Periodontal Disease; Chronic Kidney Disease
Keywords: periodontal disease; CKD; nutrition; inflammation; anemia response to ESA; quality of life; hemodialysis
MeSH Terms: conditions — Periodontal Diseases; Renal Insufficiency, Chronic; Inflammation | interventions — Dental Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Dental treatment: Assessment of the clinical state of the patient. Professional prophylaxis and removal of calculus. Extraction of hopeless teeth.Education of patient for oral hygiene. Periodic reevaluation.
  Interventions: Other: Dental treatment

INTERVENTIONS:
Other: Dental treatment — 1. The preliminary stage deals with:
     * assessment of the clinical state of the patient by completing a detailed dental and periodontal chart
     * education of the patient regarding correct oral hygiene habits;
  2. Phase I Therapy:
     * plaque control : removal of dental plaque, calculus and root planning; antimicrobial therapy (local or systemic)
     * evaluation of response to the treatment
  3. Phase II Therapy - surgical phase:
     * extraction of hopeless teeth
     * evaluation of the surgical results.
  4. Maintenance phase:
     * periodic reevaluation of plaque and calculus and of periodontal conditions.

SUMMARY:
Several studies revealed a direct relationship between the severity of periodontal inflammation and CRP (NHANES III, Dumitriu HT et al, 1998). In patients without any other source of inflammation but PDD, proper dental treatment of the disease decreased CRP to normal levels (Dumitriu H.T. et al., 1998; D'Aiuto F. et al, 2004; Borawski J. et al., 2007) Moreover, a direct link between high levels of CRP and atherosclerotic complications has been found in studies conducted both in general population (Ridker PM, et al., 1998; Koenig W, et al., 1999) and in HD subjects (Westhuyzen J, et al., 2000; Iseki K., et al., 1999; Zimmermann J, et al. 1998).

DETAILED DESCRIPTION:
Patients will be recruited according to eligibility criteria. Initial oral and general status will be evaluated and recorded. The evaluated parameters are listed at the study description section. Also, quality of life will be assessed by using the SF-36 and OHIP-14 questionnaires.

Patients will undergo a series of dental interventions with the final scope of eliminating all oral inflammation. Participants will also be instructed regarding correct oral hygiene habits.

Following dental and periodontal treatments, the oral and general status will be reassessed and the obtained dat analysed.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialyzed patients with periodontal disease

Exclusion Criteria:

* Malignancies, Diabetes
* Patient refusal to participate

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Haemodialyzed patients with Periodontal Disease
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-09 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Modification of nutritional status | 6 months
  SGA, whole body bioimpedance, biochemical parameters (serum albumin, predialysis serum urea, serum creatinine, serum phosphates)

SECONDARY OUTCOMES:
Modification of inflammatory status | 6 months
  C Reactive Protein

OTHER OUTCOMES:
Modification of periodontal disease index | 3 months
  Modification of periodontal disease index assessed by the CAL, PPD, bleeding index
Modification of the quality of life, as assessed by SF-36 and OHIP-14 | 6 months
  Modification of the quality of life, as assessed by SF-36 and OHIP-14
Modification of anaemia response to epoetin | 6 months
  Modification of anaemia response to epoetin, as assessed by the ERI and by the cumulative ESAs dose

CONTACTS AND LOCATIONS:
Overall Officials: Oana Slusanschi, DMD, Principal Investigator — University of Medicine and Pharmacy Bucharest
Locations (1):
- CMI "Dr Slusanschi Oana", Bucharest, Romania